CLINICAL TRIAL: NCT03909035
Title: Medication Reviews Performed for Elderly Patients: a Collaborative Approach Between Community Pharmacists, Patients and General Practitioners to the Optimizations of Prescriptions
Brief Title: A Collaborative Approach to Medication Reviews for Older Patients With Polypharmacy
Acronym: BIMEDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/17/0454; 17-0277 (Other Grant/Funding Number: French Ministry of Health, PREPS 2017); 2018/A00213/52 (Other: ANSM)
Record Dates: First submitted 2019-03-19; First posted 2019-04-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Medication Therapy Management
Keywords: Medication review polypharmacy; clinical pharmacy; older people; inappropriate prescribing; collaboration
MeSH Terms: interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication therapy management (Experimental): Medication therapy management by the community pharmacist in collaboration with the General Practitioners to the Optimizations of Prescriptions
  Interventions: Other: Medication therapy management
- Usual pharmaceutical care (No Intervention): Usual pharmaceutical care provided by the community pharmacist (first level pharmaceutical analysis of the prescriptions)

INTERVENTIONS:
Other: Medication therapy management — The intervention is in the form of a pharmacist-led medication review aimed at detecting potentially inappropriate prescribing. It includes:
  * A patient-pharmacist interview to collect comorbidities, medication, laboratory results, self-medication, adherence, medication patient's knowledge.
  * A pharmacist's evaluation of the prescriptions based on the patient's conditions and on the current recommendations for clinical practice.
  * Detailed feedback to the general practitioner.
  * An appointment with the patient to explain the modifications made by the general practitioner (GP)
  Arms: Medication therapy management

SUMMARY:
In patients aged 65 years and older, polypathology is frequent and often associated with polypharmacy. This polypharmacy may be a source of iatrogeny due to pharmacokinetic interactions, enhanced sensitivity of older people to medication, or failure to adhere to the therapy. Since January 2018, French community pharmacists have been allowed by the Health ministry to perform medication reviews for people aged 65 years and over, who are being treated with more than 5 medications a day. the present hypothesis is that medication therapy management performed in collaboration with patients, general practitioners, and community pharmacists will lead to a reduction in medical events and inappropriate prescriptions.

DETAILED DESCRIPTION:
This is a stepped-wedge cluster randomised controlled trial conducted in 9 regions of France. Each region represents one cluster with 7 community pharmacies located around the University Hospital associated with that cluster. In total, 63 community pharmacies will be enrolled, with each pharmacy including 20 patients over a 10 month-period. Over the life-time of the project, a total of 1260 patients will benefit from either the intervention or from a controlled pharmaceutical care according to the period of time they will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 65 or older suffering from long-term illness
* Patient aged 75 or older
* Living at home
* Having 5 medications or more per day for more than 6 months
* Being a regular patient of the community pharmacy involved in the study
* General practitioner of the patient agrees to participate to the study
* Patient being mentally and physically able to decide on his own to participate in the study
* Patient available by phone throughout the study

Exclusion Criteria:

* Patient refuses to participate
* Patient without a family doctor
* Patient whose family doctor refuses to participate in the study
* Patient who does not understand French, or dependant on someone else to manage his medication
* Resident of a nursing home
* Patient placed under guardianship
* Uncertainty of the pharmacist about patient reliability
* Patient having benefited from a medication review in the previous 12 months
* Patient already included in another study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 697 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Number of patients hospitalised | Month 12
  Number of patients hospitalised for more or less than 24 hours, including emergency department transfers during a 12 month-period follow-up.

SECONDARY OUTCOMES:
Number of patients hospitalised (only non-scheduled hospitalisations) | Month 12
  Number of non-scheduled hospitalisations (including emergency department transfers)
Existence of at least one potentially inappropriate drug per patient | Month 0
  Evolution of potentially inappropriate prescribing
Existence of at least one potentially inappropriate drug per patient | Month 2
  Evolution of potentially inappropriate prescribing
Existence of at least one potentially inappropriate drug per patient | Month 12
  Evolution of potentially inappropriate prescribing
Mean number of medications per patient | Month 0
  Mean number of medications per patient
Mean number of medications per patient | Month 12
  Mean number of medications per patient
Medication regimen complexity index | Month 0
  Medication regimen complexity index
Medication regimen complexity index | Month 12
  Medication regimen complexity index
Girerd compliance test score | Month 0
  To evaluate the impact of medication therapy management on Medication adherence. From 0 to 6 Yes. 0 Yes: Best value. 6 Yes: worst value.
Girerd compliance test score | Month 4
  To evaluate the impact of medication therapy management on Medication adherence.From 0 to 6 Yes. 0 Yes: Best value. 6 Yes: worst value.
  From 0 to 6 Yes. 0 Yes: Best value. 6 Yes: worst value.
Girerd compliance test score | Month 8
  To evaluate the impact of medication therapy management on Medication adherence. From 0 to 6 Yes. 0 Yes: Best value. 6 Yes: worst value.
Girerd compliance test score | Month 12
  To evaluate the impact of medication therapy management on Medication adherence. From 0 to 6 Yes. 0 Yes: Best value. 6 Yes: worst value.
Quality of life measured with the EuroQol Group 5-level EQ-5D version | Month 0
  To evaluate the impact of medication therapy management on The patients' quality of life: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Quality of life measured with the EuroQol Group 5-level EQ-5D version | Month 4
  To evaluate the impact of medication therapy management on The patients' quality of life: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Quality of life measured with the EuroQol Group 5-level EQ-5D version | Month 8
  To evaluate the impact of medication therapy management on The patients' quality of life: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Quality of life measured with the EuroQol Group 5-level EQ-5D version | Month 12
  To evaluate the impact of medication therapy management on The patients' quality of life: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Differential cost ratio | Month 4
  To evaluate the impact of medication therapy management on The cost-utility and cost-efficacy ratios
Differential cost ratio | Month 8
  To evaluate the impact of medication therapy management on The cost-utility and cost-efficacy ratios
Differential cost ratio | Month 12
  To evaluate the impact of medication therapy management on The cost-utility and cost-efficacy ratios
Mean number of modifications made by the General Practitioner per patient, following the pharmacist's intervention | Month 2
  To evaluate the modifications made by the general practitioner due to the pharmacists' interventions

CONTACTS AND LOCATIONS:
Overall Officials: Cestac, Principal Investigator — Toulouse University Hospital / Paul Sabatier University
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No